CLINICAL TRIAL: NCT04679272
Title: Prognostic Evaluation of COVID-19 in Rheumatoid Arthritis Patients : ProCOVRA
Brief Title: Prognostic Evaluation of COVID-19 in Rheumatoid Arthritis Patients
Acronym: ProCOVRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0682
Record Dates: First submitted 2020-12-20; First posted 2020-12-22 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Rheumatoid Arthritis
Keywords: DMARDs; Biotherapy
MeSH Terms: conditions — COVID-19; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is an infectious disease caused by SARS-CoV2 virus. The objective of our study is to analyze the progression and the severity of COVID-19 in patients with RA. Indeed, few data are available on this subject, and this would allow us to improve management of COVID-19 in these potential at-risk patients.

ELIGIBILITY:
Inclusion criteria:

- Confirmed COVID-19 diagnosis (positive PCR or serology) in RA patients or healthy controls.

Exclusion criteria:

* Age under 18 years old
* Suspected COVID-19 diagnosis (typical symptoms without a positive PCR or serology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population description: *
  * Patients with RA, included in the French RMD Covid-19 cohort, with a confirmed COVID-19 diagnosis (positive PCR or serology).
  * Patients included in the Montpellier COVID-19 cohort, without autoimmune disease or inflammatory rheumatism, and with a confirmed COVID-19 diagnosis (positive PCR or serology).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization rates for COVID-19 | 1 day
  Proportion of hospitalized patients in RA group or control group. From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.

SECONDARY OUTCOMES:
Critical care transfer rate for COVID-19 and death due to COVID-19 | 1 day
  Proportion of patients transferred in critical care for COVID-19 or deaths due to COVID-19 From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.
Pulmonary comorbidities, corticosteroids or DMARDs use | 1 day
  Type and severity of patients pulmonary comorbidities and treatment by corticosteroids or DMARDs in RA group From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.
Age | 1 day
  Patients demographics From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.
Number of Participants with co-morbidities | 1 day
  Patients comorbidities From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.
Type of clinical presentation | 1 day
  Patients COVID-19 clinical presentation From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.
Type of associated treatments | 1 day
  From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Padern Guillaume, physician, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC